CLINICAL TRIAL: NCT00181584
Title: Zoledronic Acid to Prevent Bone Loss During Androgen Deprivation Therapy for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Matthew R. Smith, MD, PhD, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 03-194
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Bone Loss; Prostate Cancer
Keywords: Androgen deprivation therapy; bone loss; prostate cancer; Zoledronic Acid; Zometa
MeSH Terms: conditions — Bone Diseases, Metabolic; Prostatic Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Drug: Zoledronic acid
- Group 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Zoledronic acid — Given intravenously once.
  Other Names: Zometa
  Arms: Group 1
Other: Placebo — Given intravenously once.
  Arms: Group 2

SUMMARY:
The primary objective of this study is to determine whether zoledronic acid (Zometa) given once annually increases bone mineral density in men receiving hormone therapy for prostate cancer.

DETAILED DESCRIPTION:
* Patients will be randomized into 2 groups. At the screening visit, a bone mineral density test will be performed to determine if the patient has osteoporosis or not. Patients with osteoporosis will be treated with Zometa. Patients without osteoporosis will be randomly assigned to receive either Zometa or a placebo.
* Zometa is administered intravenously over a 15 minute prior once in this one year study.
* All patients will asked to take an over-the-counter oral calcium (500mg daily) and a daily multi-vitamin (containing 400-500 I.U of vitamin D) during the study.
* All patients will have clinic visits every 3 months for blood tests and to report any side effects they may be experiencing. At month 12, a bone mineral density test will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate
* Current androgen deprivation therapy with expected duration of treatment greater than or equal to 12 months
* Corrected serum calcium > 8.4mg/dl and < 10.6mg/dl
* Serum creatinine < 2.0mg/dl

Exclusion Criteria:

* History of bone metastases by bone scan
* Treatment with bisphosphonate within one year
* History of metabolic disease
* Chronic use of glucocorticoids, anticonvulsants, or suppressive doses of thyroxine within one year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-09; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
To compare change in bone mineral density from baseline to one year between men treated with Zometa (zoledronic acid) and men treated with placebo. | 3 years

SECONDARY OUTCOMES:
To compare changes in biochemical markers of bone turnover between men treated with zoledronic acid and men treated with placebo | 3 years
to assess the safety and tolerability of zoledronic acid. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Smith, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts